CLINICAL TRIAL: NCT01868269
Title: Multinational European Trial for Children With the Opsoclonus Myoclonus Syndrome / Dancing Eye Syndrome
Brief Title: Opsoclonus Myoclonus Syndrome/Dancing Eye Syndrome (OMS/DES) in Children With and Without Neuroblastoma (NBpos and NBneg)Opsoclonus Myoclonus Syndrome/Dancing Eye Syndrome (OMS/DES) in Children With and Without Neuroblastoma (NBpos and NBneg)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2011-02
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Opsoclonus Myoclonus Syndrome; Neuroblastoma
MeSH Terms: conditions — Opsoclonus-Myoclonus Syndrome; Neuroblastoma | interventions — dexamethasone acetate; Dexamethasone; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexamethasone Cyclophosphamide Rituximab (Other)
  Interventions: Drug: Dexamethasone acetate; Drug: dexamethasone and cyclophosphamide; Drug: dexamethasone and rituximab

INTERVENTIONS:
Drug: Dexamethasone acetate — First step:
  immunosuppressive treatment with dexamethasone
Drug: dexamethasone and cyclophosphamide — second step (in case of insufficient response): immunosuppressive treatment with dexamethasone and cyclophosphamide
Drug: dexamethasone and rituximab — third step (in case of insufficient response): immunosuppressive treatment with dexamethasone and rituximab

SUMMARY:
The OMS/DES study is a multinational European Trial for Children with the Opsoclonus Myoclonus Syndrome / Dancing Eye Syndrome.

This trial brought on the way by specialists of the EPNS (European Paediatric Neurology Society), the GPOH (Gesellschaft für Pädiatrische Hematologic und Oncologie) and the SIOPEN (SIOP (International Society Oncology Pediatric) Europe Neuroblastoma).

This protocol will investigate an escalating treatment schedule starting with a corticosteroid standard treatment with dexamethasone pulses (first step), which is followed, if response has been inadequate after 3 months of treatment, by the addition of CP (second step) and, if still no sufficient improvement, by the replacement of CP by Rituximab (third step). Treatment intensification is decided on the basis of standardized scoring of OMS/DES severity.

ELIGIBILITY:
Inclusion Criteria:

* Children with newly diagnosed OMS/DES either NB-pos or NB-neg.

Three out of the following four components are necessary for the diagnosis of OMS/DES:

* Opsoclonus or ocular flutter (but not nystagmus)
* Ataxia and/or myoclonus
* Behavioural change and/or sleep disturbance
* Neuroblastoma The diagnosis of OMS/DES may be difficult in some patients. Opsoclonus, in particular, may be intermittent or late in onset. A video example will be available at www.dancingeyes.org.uk. If uncertain, please contact the national coordinator for support in interpreting clinical features.

  * Age 6 months or over up to less than 8 years (< 8th birthday) The date of diagnosis of OMS/DES is the date on which a doctor confirms the condition to be OMS/DES. The date of symptom onset needs also to be documented.
  * Treatment start with the standard corticosteroid treatment with dexamethasone pulses as proposed by the guidelines given in this trial protocol (see 11.10, page 71).
  * In patients with presumed NB-neg OMS/DES, neuroblastoma must be excluded according the guidelines of this trial (see chapter 4.4.1.4, page 30, and appendix 11.9, page 70)
  * Documented informed consent for treatment and enrolment in the trial by parents / legal representatives.

Exclusion Criteria:

•Patients with opsoclonus, myoclonus or ataxia caused by other identified disease (e.g. current active CNS infection, neurometabolic disorder or demyelination).

An identified viral precursor is not an exclusion criterion.

* prior or parallel use of chemotherapy (other than required for treatment of the neuroblastoma)
* Corticoid steroid for OMS/DES or other reasons lasting 14 days or more immediately before treatment start according the standard treatment proposed (treatment with corticosteroids for less than 14 days will be allowed)
* contre-indication of use of one of the experimental study drug (cf Summary of Product Characteristics used in this study)

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
The response to treatment schedule as defined by the percentage of patients with disappearance of all symptoms. | at 48 weeks after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Schleiermacher, MD, Principal Investigator — Institut Curie
Locations (36):
- St. Anna Kinderkrebsforschung e.V. CHILDREN'S CANCER RESEARCH INSTITUTE, Vienna, Austria
- France (29):
  - Chu de Bicetre, Le Kremlin-Bicêtre, LE Kremlin Bicetre
  - Centre Oscar Lambret, Lille, Lille Cedex
  - Centre Leon Berard, Lyon, LYON Cedex 08
  - Hopita D'Enfants de La Timone, Marseille, Marseille Cedex 5
  - Hopital Arnaud de Villeneuve, Montpellier, Montpellier Cedex 4
  - Chr de Nantes, Nantes, Nantes Cedex01
  - Chu de Nice Archet 2, Nice, NICE Cedex 03
  - Ch Trousseau, Paris, Paris Cedex 12
  - Chu Hopital Sud, Rennes, Rennes Cedex 02
  - Chu de Rouen, Rouen, Rouen Cedex
  - CHU DE STRASBOURG HOPITAL Hautepierre, Strasbourg, Strasbourg Cedex
  - Chu Toulouse Hopital Des Enfants, Toulouse, Toulouse Cedex 9
  - Chu Amiens, Amiens
  - Chu Angers, Angers
  - Hopital Jean Minjoz, Besançon
  - Chr Pellegrin, Bordeaux
  - CHU CAEN, Caen
  - Chu D'Estaing, Clermont-Ferrand
  - Chu Dijon, Dijon
  - Chu de Grenoble, Grenoble
  - Chu de Limoges, Limoges
  - Institut Curie, Paris
  - Chu de Poitiers, Poitiers
  - Chu de Reims, Reims
  - CHU LA REUNION Site Félix Guyon, Saint-Denis
  - Chu Saint Etienne, Saint-Etienne
  - Chu Tours Hopital Clocheville, Tours
  - Hopital Nancy Brabois, Vandœuvre-lès-Nancy
  - Institut de Cancerologie Gustave Roussy, Villejuif
- G. Gaslini Institut, Genova, Italy
- The Fundación para la Formación e Investigación Sanitarias de la Región de Murcia, El Palmar, Spain
- University Hospital Lund, Lund, Sweden
- Switzerland (2):
  - Universitätskinderklinik, Bern
  - Kinderspital Zurich, Zurich
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).